CLINICAL TRIAL: NCT04222504
Title: Community-based Venues for Delivery of Healthcare Services in Umlazi, South Africa: Proof of Concept Pilot Conducted in Hair Salons
Brief Title: Community-based Venues for Delivery of Healthcare Services: Proof of Concept Pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Adrenergy Research Innovations (Unknown)
Responsible Party: Principal Investigator, Ingrid V. Bassett, MD, MPH, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019P003869; K24AI141036 (NIH); BFC449/19 (Other: UKZN Biomedical Research Ethics Committee)
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pre-Exposure Prophylaxis; STI; Contraceptive Usage
MeSH Terms: conditions — Sexually Transmitted Diseases; Contraception Behavior | interventions — Emtricitabine; Hormonal Contraception; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Salons (Experimental): Intervention: Behavioral: Provision of sexual health preventative services in the salon setting
  Interventions: Behavioral: Provision of sexual health preventative services in the salon setting
- Control Salon (No Intervention): No Intervention

INTERVENTIONS:
Behavioral: Provision of sexual health preventative services in the salon setting — Participants at intervention salons will be offered a choice of receiving daily PrEP and/or contraceptives (oral and injectables). Participants that elect to receive at least PrEP or contraceptives will also be offered STI testing.
  Follow-up visits will be planned for 3, 6, 9, and 12-months. Attendance at follow-up visits for monitoring and medication refill will be encouraged using text message reminders, WhatsApp support groups, and lottery-based incentives for free salon services.
  Other Names: PrEP (combined tenofovir/emtricitabine); STI testing; Hormonal birth control (Oral, Injectable)
  Arms: Intervention Salons

SUMMARY:
The investigators propose to offer a package of evidence-based health services to women in two hair salons in the Umlazi township of Durban. Based on community feedback in previous survey and qualitative work, the package has been designed to include daily PrEP, family planning/contraceptives, and STI screening. Interested salon clients at intervention salons will elect which services to use. An additional salon will serve as control, offering no health services to clients. Surveys will be conducted in both salon groups. Attendance at follow-up visits for monitoring and medication refill will be encouraged using text message reminders, WhatsApp support groups, and lottery-based incentives for free salon services. Recruitment in intervention salons will conclude when 100 clients uptake PrEP, not inclusive of clients who enroll at intervention salons who accept other services through the study. Approximately 250 participants will be recruited in control salons. The study team anticipates an overall total enrollment of 500.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years or older
* English or Zulu speaking
* Able and willing to consent

Exclusion Criteria:

* Symptoms of acute HIV viral syndrome
* Known pregnancy at baseline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of Preventative Sexual Health Services | Months 4 to 16
  We will measure uptake of the intervention as the proportion of eligible women who agree to salon-based contraception (first-time users and new users) and separately to salon-based PrEP.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid V. Bassett, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Adrenergy Research Innovations, Durban, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jarolimova J, Yan J, Govere S, Shezi S, Ngcobo LM, Sagar S, Zionts D, Dube N, Parker RA, Bassett IV. Sexually Transmitted Infection Testing Integrated With HIV Prevention and Contraceptive Services in Hair Salons in Urban South Africa. J Acquir Immune Defic Syndr. 2025 Aug 1;99(4):359-367. doi: 10.1097/QAI.0000000000003677. PMID 40192662
- [Derived] Bassett IV, Yan J, Govere S, Shezi S, Ngcobo LM, Sagar S, Jarolimova J, Zionts D, Khumalo A, Zwane Z, Psaros C, Dube N, Parker RA. A pilot cluster randomized controlled trial assessing uptake of PrEP and contraception in hair salons in South Africa. BMC Public Health. 2025 Feb 8;25(1):524. doi: 10.1186/s12889-025-21718-3. PMID 39922997
- [Derived] Govere SM, Jarolimova J, Yan J, Shezi S, Ngcobo LM, Sagar S, Zionts D, Dube N, Parker RA, Psaros C, Bassett I. Uptake of HIV pre-exposure prophylaxis and contraception in South African hair salons: a study protocol for a pilot cluster randomised controlled trial. BMJ Open. 2024 Dec 20;14(12):e083621. doi: 10.1136/bmjopen-2023-083621. PMID 39806604